CLINICAL TRIAL: NCT00602446
Title: Open-Label Single-Arm Pilot Study of Deferasirox (Exjade®) in Adult Allogeneic Hematopoietic Stem Cell Transplant Recipients With Transfusional Iron Overload
Brief Title: Deferasirox in Treating Patients With Iron Overload After Undergoing a Donor Stem Cell Transplant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow accrual of patients
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000584690; UMN-2007LS065 (Other: Masonic Cancer Center, University of Minnesota); UMN-MT2007-11R (Other: Blood and Marrow Transplantation Program); NOVARTIS-CICL670AUS12 (Other: Novartis Pharmaceuticals)
Record Dates: First submitted 2008-01-24; First posted 2008-01-28 (Estimated); Results first posted 2010-03-30 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer; Iron Overload; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Neuroblastoma; Ovarian Cancer
Keywords: iron overload
MeSH Terms: conditions — Breast Neoplasms; Iron Overload; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Neuroblastoma; Ovarian Neoplasms | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Deferasirox Treated (Experimental): Includes patients that were treated with deferasirox for 6 months.
  Interventions: Drug: deferasirox

INTERVENTIONS:
Drug: deferasirox — 20 mg/kg once daily orally for 6 months
  Other Names: Exjade

SUMMARY:
RATIONALE: Deferasirox may be effective in treating iron overload caused by blood transfusions in patients who have undergone donor stem cell transplant.

PURPOSE: This phase II trial is studying the side effects and how well deferasirox works in treating patients with iron overload after donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the safety of deferasirox given over 6 months in reducing liver iron concentration in patients with transfusional iron overload after undergoing allogeneic hematopoietic stem cell transplantation.

Secondary

* To evaluate the efficacy of deferasirox in reducing liver iron overload in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral deferasirox once daily for 6 months in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of iron overload, defined as serum ferritin > 1,000 ng/mL and liver iron concentration ≥ 5 mg iron/g on tissue proton transverse relaxation rates Magnetic Resonance Imaging (MRI)
* Underwent prior allogeneic hematopoietic stem cell transplantation (HSCT) using either myeloablative or reduced-intensity conditioning at least 12 months ago
* No evidence of relapse or progression of the primary disease for which allogeneic HSCT was performed
* Patients who have become red-cell transfusion independent (i.e., no red cell transfusions within the past 3 months) as well as patients who require red cell transfusions are eligible
* Meets one of the following criteria:

  * Ineligible for phlebotomy (hemoglobin < 11 g/dL, poor intravenous access, or unable to undergo phlebotomy every 4 weeks)
  * Have failed treatment with phlebotomy (serum ferritin > 50% of baseline after 3 months of phlebotomy)
  * Refused phlebotomy
* ECOG performance status of 0-2
* Life expectancy ≥ 6 months
* Adequate renal function defined as serum creatinine < or = 1.6 mg/dL and creatinine clearance of > or = 60 ml/min calculated using the Crockcroft-Gault formula on 2 occasions within 30 days of enrollment
* Sexually active men and women must use an effective method of contraception. Alternatively, women must have undergone clinically documented total hysterectomy and/or oophorectomy, or tubal ligation or be postmenopausal.
* Must be able to give written informed consent.
* Prior therapy with deferoxamine allowed provided it was completed ≥ 12 months ago

Exclusion Criteria:

* Contraindication for performing MRI or inability to undergo MRI because of claustrophobia or weight (>350 pounds).
* Inability to take medications orally.
* Uncontrolled bacterial, viral, or fungal infection
* ANC ≥ 1,000/mm³
* Hemoglobin ≥ 8.0 g/dL
* Platelet count ≥ 50,000/mm³
* Aspartate aminotransferance (AST) and alanine aminotransferase (ALT) ≤ 5 times the upper limit of normal
* Less than 4 weeks since prior and no concurrent systemic investigational drug
* Less than 7 days since prior and no concurrent topical investigational drug. Concurrent non-investigational medications needed to treat concomitant medical conditions are allowed, with the exception of other chelating agents. Concurrent growth factors such as epoetin alfa, darbepoetin alfa, filgrastim (G-CSF), and sargramostim (GM-CSF) allowed. Concurrent irradiated packed red-cell and platelet transfusions allowed as clinically indicated. Concurrent low-doses of vitamin C supplements (≤ 200 mg/day) allowed.
* Concurrent iron supplements or multivitamins with iron.
* Aluminum-containing antacid therapies may not be taken simultaneously with deferasirox, but may be taken 2 hours before or after administration of deferasirox
* On dialysis or status post-renal transplantation
* Pregnant or nursing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-08; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda J. Burns, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only one site (Masonic Cancer Center) enrolled patients in this study.
Pre-assignment Details: 4 patients were consented, however, one withdrew consent before receiving treatment.
Period: Overall Study
Arm/Group | Deferasirox Treated
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Deferasirox Treated
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Not Completing Treatment
Description: Number of patients who discontinued deferasirox during 6 month daily treatment due to drug related toxicity
Time Frame: 6 Months
Population: Note: 1 patient had a transient decrease in hemoglobin that required discontinuation of treatment for 2 weeks; subsequently restarted at same dose and completed therapy.
Measure: Number; unit: Participants
Arm/Group | Deferasirox Treated
Number analyzed (Participants) | 3
Participants | 0

2. Secondary Outcome: Reduction in Liver Iron Concentration After Study Drug
Description: Efficacy as measured by reduction in liver iron concentration (LIC) after 6 months of the study drug compared to baseline (LIC at baseline minus LIC at 6 months). This shows the mean reduction for the 3 subjects treated in this study.
Time Frame: 6 Months
Population: All patients included in count.
Measure: Mean (Standard Deviation); unit: milligrams/gram
Arm/Group | Deferasirox Treated
Number analyzed (Participants) | 3
milligrams/gram | 5.6 (4.8)

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Deferasirox Treated
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferasirox Treated (N=3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Increased serum creatinine (Blood and lymphatic system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No